CLINICAL TRIAL: NCT04718740
Title: A Phase I, Multi-center Study to Determine the Effect of Fluzoparib on Pharmacokinetics of Caffeine, S-Warfarin, Omeprazole, Midazolam, Repaglinide and Bupropion in Patients With Recurrent Ovarian Cancer
Brief Title: A Drug-drug Interaction Study Of Fluzoparib (SHR3162) on Patients With Recurrent Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: FZPL-Ⅰ-120
Record Dates: First submitted 2021-01-14; First posted 2021-01-22 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Recurrent Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — fluzoparib; Caffeine; Vitamin K; Warfarin; Omeprazole; Midazolam; repaglinide; Bupropion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- fluzoparib (Experimental): * Experimental: group A Intervention: Drug: fluzoparib, caffeine, vitamin K, warfarin, omeprazole, and midazolam
  * Experimental: group B Intervention: Drug: fluzoparib, repaglinide and bupropion
  Interventions: Drug: fluzoparib

INTERVENTIONS:
Drug: fluzoparib — Group A: Caffeine, vitamin K, warfarin, omeprazole, and midazolam with or without fluzoparib Group B: Repaglinide and bupropion with or without fluzoparib
  Other Names: caffeine, vitamin K, warfarin, omeprazole, midazolam, repaglinide and bupropion

SUMMARY:
Primary objective: To evaluate the pharmacokinetic effects of fluzoparib on caffeine, S-warfarin, omeprazole, midazolam, repaglinide and bupropion in patients with recurrent ovarian cancer.

Secondary objective: To evaluate the safety of single dose of fluzoparib, caffeine, S-warfarin, omeprazole, midazolam, repaglinide and bupropion or fluzoparib in combination with caffeine, S-warfarin, omeprazole, midazolam, repaglinide and bupropion in patients with recurrent ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to enter the study:

1. Patients are willing to participate this research and sign informed consent forms (ICFs)
2. Patients must be ≥ 18 years of age at the date of signing the informed consent;
3. Patients with histologically diagnosed relapsed high grade (or middle and low differentiation) serous ovarian cancer, fallopian tube cancer or primary peritoneal cancer confirmed by pathology; ovarian endometrioid adenocarcinoma ≥ grade II; mixed type tumor: high grade serous type or endometrioid component ≥ grade II should be more than 50%;
4. Patients with platinum sensitive recurrent ovarian cancer, fallopian tube cancer or primary peritoneal cancer achieved complete or partial remission after platinum containing chemotherapy (carboplatin and cisplatin only). Platinum sensitive defined as having disease progression greater than 6 months after completion of their last dose of platinum chemotherapy. Patient must have received, at least 4 cycles of a platinum based chemotherapy regimen for the last chemotherapy course
5. ECOG Performance Status of 0-1
6. Patients must have a life expectancy of at least 3 months
7. Patients must have normal organ and bone marrow function measured prior to administration of study treatment as defined below:

   HB≥100g/L； ANC≥1.5×109/L； PLT≥100×109/L or 1x UN TBIL≤1.5×ULN； ALT和AST≤3×ULN； Cr≤1.5×ULN； Albumin>30g/L；
8. Agree to abstain from sex or use effective non-drug contraceptives from screening to at least 6 months after the last study drug administration (female subjects are also required to abstain or use effective non-drug contraceptives two weeks prior to study entry)

Exclusion Criteria:

Inclusion Criteria:

Subjects must meet all of the following criteria to enter the study:

1. Patients are willing to participate this research and sign informed consent forms (ICFs)
2. Patients must be ≥ 18 years of age at the date of signing the informed consent;
3. Patients with histologically diagnosed relapsed high grade (or middle and low differentiation) serous ovarian cancer, fallopian tube cancer or primary peritoneal cancer confirmed by pathology; ovarian endometrioid adenocarcinoma ≥ grade II; mixed type tumor: high grade serous type or endometrioid component ≥ grade II should be more than 50%;
4. Patients with platinum sensitive recurrent ovarian cancer, fallopian tube cancer or primary peritoneal cancer achieved complete or partial remission after platinum containing chemotherapy (carboplatin and cisplatin only). Platinum sensitive defined as having disease progression greater than 6 months after completion of their last dose of platinum chemotherapy. Patient must have received, at least 4 cycles of a platinum based chemotherapy regimen for the last chemotherapy course
5. ECOG Performance Status of 0-1
6. Patients must have a life expectancy of at least 3 months
7. Patients must have normal organ and bone marrow function measured prior to administration of study treatment as defined below:

   HB≥100g/L； ANC≥1.5×109/L； PLT≥100×109/L or 1x UN TBIL≤1.5×ULN； ALT和AST≤3×ULN； Cr≤1.5×ULN； Albumin>30g/L；
8. Agree to abstain from sex or use effective non-drug contraceptives from screening to at least 6 months after the last study drug administration (female subjects are also required to abstain or use effective non-drug contraceptives two weeks prior to study entry)

Exclusion Criteria:

Subjects who do meet any of the following criteria will not be allowed to enter the study:

1. Patients with previously (within 5 years) or at the same time with other incurable malignant tumors, except for cured skin basal cell carcinoma, cervical carcinoma in situ and breast cancer with no recurrence for more than 5 years after radical operation
2. 3 months prior treatment with any poly adenosine diphosphate ribose polymerase inhibitor (PARPi)
3. Patients with central nervous system metastasis
4. Serous cavity effusion (including pleural effusion, ascites and pericardial effusion) with clinical symptoms and requiring symptomatic treatment; note: Patients with symptomatic serous cavity effusion can be included in the group if there is no disease, patients with symptomatic serous cavity effusion can be included in the group if they are treated with symptomatic treatment (anti-cancer drugs can not be used for serous cavity effusion treatment), and patients can be included in the group if judged by researchers
5. Pre-existing duodenal stent, recent or existing bowel obstruction, and/or any gastrointestinal disorder or defect that would interfere with absorption of study drugs
6. There are clinical cardiac symptoms or diseases that can not be well controlled, such as: (1) NYHA grade 2 or above cardiac insufficiency, (2) unstable angina pectoris, (3) acute myocardial infarction within one year, (4) clinically significant supraventricular or ventricular arrhythmia requiring treatment or intervention, (5) QTc > 470ms
7. Patients with abnormal coagulation function (INR > 1.5 or PT > ULN + 4 seconds), bleeding tendency or receiving thrombolytic or anticoagulant therapy
8. Contraindications of midazolam (allergic to benzodiazepine, myasthenia gravis, schizophrenia, severe depression patients)
9. Warfarin contraindications (liver and kidney dysfunction, severe hypertension, coagulation dysfunction with bleeding tendency, active ulcer, trauma, threatened abortion, recent surgery)
10. Patients with contraindications to repaglinide and bupropion (patients with type I diabetes, including insulin-dependent IDDM and C-peptide negative diabetes, diabetic ketoacidosis with or without coma, patients with anorexia nervosa or bulimia, patients with a history of severe epilepsy; patients with sudden abstinence or withdrawal of sedatives); patients with diabetes other than the above Abnormal control
11. Not recovered from the previous adverse events before the first medication (previous treatment adverse events, excluding hair loss and fatigue, recovered to ≤ 1 level)
12. Other clinical trial drugs were taken within 4 weeks before the first medication;
13. CYP1A2, CYP3A4, CYP2C9, CYP2C19 inducers or CYP1A2, CYP3A4, CYP2C9 and CYP2C19 inhibitors or P-gp inhibitors were taken within 4 weeks before the first medication (for group A); CYP3A4, cyp2c8 and CYP2B6 inducers were taken within 4 weeks before the first medication or CYP3A4, cyp2c8 and CYP2B6 inhibitors or transporter OATP1B1 were taken within 2 weeks (or 5 half lives)/ P-gp inhibitor (for group B)
14. Prior treatment with chemotherapy, radiation, antibody therapy or other immunotherapy, gene therapy, vaccine therapy, angiogenesis inhibitors, or experimental drugs within 14 days prior to day 1
15. Alcoholics within 3 months before the first medication (drinking 14 units of alcohol per week: 1 unit = 285 ml of beer, or 25 ml of spirits, or 100 ml of wine), and smokers within 3 months before the first medication (smoking ≥ 5 cigarettes per day);
16. Ingestion of grapefruit or grapefruit products within 7 days before the first medication, or ingestion of food or drink containing caffeine, xanthine or alcohol within 72 hours before the first medication; strenuous exercise within 4 days before the first medication; or other factors affecting drug absorption, distribution, metabolism and excretion
17. Patients with history of immunodeficiency, including HIV positive, other acquired or congenital immunodeficiency diseases, or organ transplantation
18. Syphilis infection or active hepatitis (hepatitis B reference: HBsAg positive and HBV DNA ≥ 500 IU / ml; hepatitis C reference: HCV antibody positive and HCV copy number > upper limit of normal value)
19. Patients with active infections requiring antimicrobial therapy (e.g. antibiotics, antiviral drugs, antifungal drugs);
20. According to the judgment of the researchers, there are concomitant diseases (serious diabetes, thyroid diseases, etc.) that seriously endanger the safety of patients or affect the completion of the study
21. Patients with history of drug allergy, or allergic to apatinib or ingredients
22. The researcher judges other situations that may affect the clinical research and the judgment of research results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics parameters of caffeine, S-warfarin, omeprazole, midazolam, repaglinide, bupropion and hydroxybupropion | DAY1, DAY22
  Peak Plasma Concentration (Cmax)
Pharmacokinetics parameters of caffeine, S-warfarin, omeprazole, midazolam, repaglinide, bupropion and hydroxybupropion | DAY1, DAY22
  Area under the plasma concentration versus time curve (AUC)

SECONDARY OUTCOMES:
Pharmacokinetics parameters of caffeine, S-warfarin, omeprazole, midazolam, repaglinide, bupropion and hydroxybupropion | DAY1,DAY 22
  Half life (t1/2)
Number of Participants With Treatment-Related Adverse Events | through study completion, an average of 1 year
  Safety: Laboratory indicators, 12-lead electrocardiogram (ECG), physical examination, vital signs, adverse events (NCI-CTC AE 5.0), etc.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Wang, Ph.D., Principal Investigator — Hunan Cancer Hospitol
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided